CLINICAL TRIAL: NCT00499785
Title: Inpatient Functional and Cognitive Assessment in Older Adults With Acute Myelogenous Leukemia
Brief Title: Physical and Mental Assessment of Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000555118; CCCWFU-22A07; CCCWFU-IRB00002562
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-10

CONDITIONS: Cognitive/Functional Effects; Depression; Leukemia
Keywords: depression; cognitive/functional effects; untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Depression; Leukemia; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted with acute leukemia

SUMMARY:
RATIONALE: Learning about physical ability and mental function over time in older patients with acute myeloid leukemia may help doctors learn about the long-term effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is assessing physical and mental status in older patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Test the feasibility of pre-treatment, bedside assessment of functional and cognitive status in older adults with newly diagnosed acute myeloid leukemia (AML).

Secondary

* Obtain preliminary data regarding the predictive value of pre-treatment, bedside assessment of functional and cognitive status on overall survival, length of hospitalization and early death.

OUTLINE: This is a prospective study.

At baseline, patients complete questionnaires including the Vulnerable Elders Survey (functional status), the Mini-Mental Status Exam (cognition), and the Center for Epidemiologic Studies-Depression. Patients also undergo physical function testing via the Short Physical Performance Battery and hand grip strength. Further information parameters are obtained by periodic medical chart reviews.

Patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed newly diagnosed acute myeloid leukemia
* Planned induction chemotherapy
* Inpatient status

PATIENT CHARACTERISTICS:

* No requirement for intensive care unit support

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy for acute myeloid leukemia

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute leukemia >= 60 years of age
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
feasibility of administering a functional assessment in clinical situation | 72 hours of admission
  Assessment of physical and cognitive function via a set of physical and congnitive tests

CONTACTS AND LOCATIONS:
Overall Officials: Heidi D. Klepin, MD, Principal Investigator — Wake Forest University Health Sciences; Bayard L. Powell, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States